CLINICAL TRIAL: NCT06433856
Title: Effects of Cold Water Immersion and Percussive Gun Massage on Recovery Measures in Soccer Players
Brief Title: Neuromuscular Responses to Recovery Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Trieste (Other)
Responsible Party: Principal Investigator, Alex Buoite Stella, RTD-A, University of Trieste
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Fisioterapia1705
Record Dates: First submitted 2024-05-17; First posted 2024-05-30 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Muscle Soreness
Keywords: recovery; team sport; cryotherapy; massage guns
MeSH Terms: conditions — Myalgia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CWI (Experimental): The CWI protocol consists of participants standing, with only their underwear and a t-shirt, in a portable tub for cold water therapy (Qryo, Italy), with the water to their hips being constantly maintained at 10±0.5 °C by a cooling system that pumped and stirred the water inside the tub and around the participant's lower limbs. Water temperature and the duration of the immersion, which is 12 minutes for all the participants considering they were characterized by similar anthropometrics and body composition, were based on previous literature
  Interventions: Other: Cold Water Immersion
- PMT (Experimental): The PMT protocol is performed with the application of a percussive therapy gun (Theragun Elite, Therabody, USA). The participants rests with their underwear and a t-shirt on a treatment bed, and the percussive therapy gun with a "standard ball", 16 mm amplitude of percussions, and a frequency of 30 Hz, is applied to the thigh muscles of both lower limbs, 3 min on the anterior and 3 min on the posterior area of each thigh. The protocol is based on previous literature and adapted to the specific aims of this study.
  Interventions: Device: Percussive Massage Therapy
- PAS (No Intervention): The control condition (PAS) consists of participants resting on a chair for 12 minutes in a quiet room at 25 °C.

INTERVENTIONS:
Other: Cold Water Immersion — Cold water immersion consists in 12 min standing in 10 °C water
  Arms: CWI
Device: Percussive Massage Therapy — Percussive massage therapy is performed with a massage gun on the thigh muscles for 12 min
  Arms: PMT

SUMMARY:
Cold water immersion (CWI) and percussive massage therapy (PMT) are commonly used re-covery techniques in team sports. In particular, despite its wide use, PMT has been scarcely investigated in the literature, especially regarding neuromuscular measures and in comparison with other techniques. This study aims to evaluate and compare the acute and short-term ef-fects (24 h) of CWI and PMT on muscle strength, contractile properties, and soreness after exercise. A randomized crossover study will be performed on sixteen male soccer players (22 y, 20-27) who participate in three experimental sessions involving high-intensity training and 12-min recovery including CWI (10 °C water), bilateral PMT on the anterior and posterior thigh, or passive resting. Outcomes will be assessed immediately after the exercise protocol, after the recovery intervention, and at 24 h. Isometric knee extension (IKE) and flexion (IKF), and tensiomyography (TMG) will be assessed.Muscle soreness and fatigue will be scored from 0 to 10.

DETAILED DESCRIPTION:
Participants will be invited to participate to a cross-over randomized trial, consisting in 3 experimental sessions at 7 days of distance one from another. During each experimental session, participants will be asked to train for about 45 min at a high-intensity protocol (High-Intensity Intermittent Running, plyometric jumps and isometric chair position). After the exercise, participants will be assessed for neuromuscular function (isometric strength and tensiomyography) as well as perceived soreness and fatigue. Then, in a randomized order, participants will receive three different recovery interventions: cold water immersion, percussive massage, or a passive control condition. After the recovery intervention, outcomes are assessed again, as well as at 24 h. Isometric strength is assessed with a dynamometer during knee extension and knee flexion. Tensiomyography is performed on the thigh muscles, and time to contraction and radial displacement are considered as outcomes. Soreness and fatigue are rated by the participant from 0 to 10.

ELIGIBILITY:
Inclusion Criteria:

* being healthy
* training in soccer for more than 3 years and with a training frequency > 2 times/week

Exclusion Criteria:

* reported time-loss injuries
* using analgesics or other therapies affecting muscle function or pain

Ages: 16 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Muscle soreness | Within 10 minutes from exercise cessation (Post-Exercise); Within 10 minutes after the intervention (Post-Intervention); 24 hours from the exercise (Post-24 hours)
  Subjective evalutation of muscle soreness from 0 to 10 with a numeric rating scale (NRS), where 0 is no soreness at all, and 10 is unbearable soreness
Muscle fatigue | Within 10 minutes from exercise cessation (Post-Exercise); Within 10 minutes after the intervention (Post-Intervention); 24 hours from the exercise (Post-24 hours)
  Subjective evaluation of muscle fatigue from 0 to 10 with a numeric rating scale (NRS), where 0 is no fatigue at all, and 10 is unbearable fatigue

SECONDARY OUTCOMES:
Isometric muscle strength | Within 10 minutes from exercise cessation (Post-Exercise); Within 10 minutes after the intervention (Post-Intervention); 24 hours from the exercise (Post-24 hours)
  Isometric knee extension (IKE) and flexion (IKF) strength assessments performed on a treatment bed, with a digital handheld dynamometer
Tensiomyography | Within 10 minutes from exercise cessation (Post-Exercise); Within 10 minutes after the intervention (Post-Intervention); 24 hours from the exercise (Post-24 hours)
  Tensiomyography (TMG) will be performed on anterior and posterior thigh muscles

CONTACTS AND LOCATIONS:
Locations (1):
- CdL in Fisioterapia, Trieste, Italy

IPD SHARING:
Plan to Share IPD: No